CLINICAL TRIAL: NCT03980067
Title: Pediatric Procedural Sedation and the Relationship With Post-Discharge Negative Behavioral Changes in the Emergency Department
Brief Title: Impact of Pre-Sedation Virtual Reality Game on Post-Discharge Negative Behaviors in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Amy Drendel, Professor, DO, MS, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1300058-5
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Behavior, Child; Anxiety
Keywords: Virtual Reality; Procedural Sedation; Modified Yale Preoperative Anxiety Scale; Post-Hospitalization Behavior Questionnaire; Pediatric; Emergency Department; Ketamine
MeSH Terms: conditions — Child Behavior; Anxiety Disorders; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): The children in the experimental group will receive the standard of care (access to in room activity including television (TV) distraction if desired, parent support and distraction at bedside, and quiet time) in addition to our intervention, an interactive virtual reality game, played for a minimum of 5 minutes prior to procedural sedation.
  Interventions: Other: Virtual Reality Game
- Standard of Care (No Intervention): The children in the control group receiving standard of care will have access to in room activity including TV distraction if desired, parent support and distraction at bedside, and quiet time.

INTERVENTIONS:
Other: Virtual Reality Game — The virtual reality headset, device, and software, created by Stanford's Childhood Anxiety Reduction through Innovation and Technology (CHARIOT)program/Weightless Studio, LLC will be utilized in this study. Children in the VR intervention group will be allowed to select a distraction-based game to play with active VR content featuring interactive avatars and interactive experiences tailored to the pediatric population that allow players to do things such as control penguins sliding down a mountain while collecting pebbles for points, control puppies running in space to collect treats to the rhythm of music, and control an asteroid miner exploring an asteroid belt and collecting points based on color of asteroids collected. The game will last a minimum of 5 minutes in duration, provided participant tolerance. The participant may play longer if desired prior to receiving procedural sedation and the total length of activity played will be documented.
  Arms: Virtual Reality Group

SUMMARY:
The purpose of this study is to evaluate if a virtual reality (VR) distraction game played prior to procedural sedation for long bone fracture reduction will improve post-discharge negative behavior changes following discharge from the pediatric Emergency Department (ED).

DETAILED DESCRIPTION:
This randomized control trial will investigate the use of a virtual reality (VR) distraction game prior to IV ketamine procedural sedation for long bone fracture reduction. Prior studies have demonstrated that children undergoing anesthesia or procedural sedation can have lingering negative behavioral changes lasting several weeks after discharge home. Children who are anxious have higher rates of developing negative behavior changes. Opiate pain control and pre-operative instructional workshops have demonstrated efficacy in decreasing negative behavior outcomes. There is some evidence that distraction techniques, such as VR, can alleviate pre-procedural anxiety and pain during procedures. To our knowledge, evaluating the use of a non-pharmacologic, virtual reality intervention and its effects on reducing post-discharge negative behavior changes following discharge from the Emergency Department has not been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6 years to 17.5 years old receiving procedural sedation with IV ketamine in the Children's Hospital of Wisconsin Emergency Department for long bone fracture reduction

Exclusion Criteria:

* Moderate to severe developmental delay
* Non-English-speaking participants or parent/guardian
* Taking psychotropic medications
* History of severe motion sickness
* Currently experiencing nausea/vomiting
* History of severe visual impairment
* History of seizures
* Expected admission to the hospital post-procedure

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Post-Hospitalization Behavior Questionnaire (PHBQ) | 24 months
  Post-Hospitalization Behavior Questionnaire, a parent-report tool, with 27 items in six categories, comprising general, separation, and sleep anxieties, eating disturbance, aggression towards authority, apathy/withdrawal accesses negative behavioral changes in children post-surgery, hospitalization (Kain et al., 1996, Kain et al., 1999) or after minor ED procedures (Brodzinski et al., 2013). It takes 10 minutes and is given prior to the sedation and at 1-week via text/email, phone, or mail follow up post-discharge.
  Parents compare their child's behavior pre-hospitalization to post using the following: much less than before (1), less than before (2), same as before (3), more than before (4), and much more than before (5). Scores above 3 indicate greater maladaptive behavioral changes, below 3 indicate improvements and 3 indicates no change in behavior.

SECONDARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale (m-YPAS) | 24 months
  The m-YPAS assesses study participant's anxiety at the time of induction of anesthesia. It is completed in <1 minute, reliable, and its validity compares favorably to the State Trait Anxiety Inventory for Children (Kain, Z. 1997). The Emergency Department provider completes the m-YPAS twice during the study: on patient arrival/enrollment and immediately preceding sedation after VR intervention or standard of care.
  m-YPAS categories are activity, vocalizations, emotional expressivity, state of apparent arousal, and use of parent). Each item has Likert-type responses reflecting children behaviors and is rated from 1 to 4 or 1 to 6 (depending on the item), and higher numbers indicate the highest severity within that item.
  Scores range from 23-100 and a score >30 is defined as anxious.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Drendel, DO, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Brodzinski H, Iyer S. Behavior changes after minor emergency procedures. Pediatr Emerg Care. 2013 Oct;29(10):1098-101. doi: 10.1097/PEC.0b013e3182a5ff07. PMID 24076612
- [Background] CHARIOT Program - Childhood Anxiety Reduction through Innovation and Technology - Stanford Children's Health. (n.d.). Retrieved August 7, 2018, from https://www.stanfordchildrens.org/en/innovation/chariot
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, Nelson W, Mayes LC. Predicting which child-parent pair will benefit from parental presence during induction of anesthesia: a decision-making approach. Anesth Analg. 2006 Jan;102(1):81-4. doi: 10.1213/01.ANE.0000181100.27931.A1. PMID 16368808
- [Background] Kim JE, Jo BY, Oh HM, Choi HS, Lee Y. High anxiety, young age and long waits increase the need for preoperative sedatives in children. J Int Med Res. 2012;40(4):1381-9. doi: 10.1177/147323001204000416. PMID 22971489
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Pearce JI, Brousseau DC, Yan K, Hainsworth KR, Hoffmann RG, Drendel AL. Behavioral Changes in Children After Emergency Department Procedural Sedation. Acad Emerg Med. 2018 Mar;25(3):267-274. doi: 10.1111/acem.13332. Epub 2017 Nov 13. PMID 28992364
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Sinha M, Christopher NC, Fenn R, Reeves L. Evaluation of nonpharmacologic methods of pain and anxiety management for laceration repair in the pediatric emergency department. Pediatrics. 2006 Apr;117(4):1162-8. doi: 10.1542/peds.2005-1100. PMID 16585311
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Wismeijer AA, Vingerhoets AJ. The use of virtual reality and audiovisual eyeglass systems as adjunct analgesic techniques: a review of the literature. Ann Behav Med. 2005 Dec;30(3):268-78. doi: 10.1207/s15324796abm3003_11. PMID 16336078
- [Background] Jenkins BN, Kain ZN, Kaplan SH, Stevenson RS, Mayes LC, Guadarrama J, Fortier MA. Revisiting a measure of child postoperative recovery: development of the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery. Paediatr Anaesth. 2015 Jul;25(7):738-45. doi: 10.1111/pan.12678. Epub 2015 May 9. PMID 25958978
- [Background] Kuhlmann AYR, Lahdo N, Staals LM, van Dijk M. What are the validity and reliability of the modified Yale Preoperative Anxiety Scale-Short Form in children less than 2 years old? Paediatr Anaesth. 2019 Feb;29(2):137-143. doi: 10.1111/pan.13536. Epub 2018 Dec 23. PMID 30365208
- [Background] Thung A, Tumin D, Uffman JC, Tobias JD, Buskirk T, Garrett W, Karczewski A, Saadat H. The Utility of the Modified Yale Preoperative Anxiety Scale for Predicting Success in Pediatric Patients Undergoing MRI Without the Use of Anesthesia. J Am Coll Radiol. 2018 Sep;15(9):1232-1237. doi: 10.1016/j.jacr.2017.12.022. Epub 2018 Mar 2. PMID 29483054
- [Background] Jenkins BN, Fortier MA, Kaplan SH, Mayes LC, Kain ZN. Development of a short version of the modified Yale Preoperative Anxiety Scale. Anesth Analg. 2014 Sep;119(3):643-650. doi: 10.1213/ANE.0000000000000350. PMID 25010821

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03980067/Prot_SAP_000.pdf
  • Informed Consent Form: Consent Form (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT03980067/ICF_001.pdf
  • Informed Consent Form: Assent Form (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT03980067/ICF_002.pdf